CLINICAL TRIAL: NCT01830465
Title: Phase II Study of VELCADE in Combination With Rituximab in Patients With Relapsed or Progressed Non Hodgkin's Follicular Lymphoma
Brief Title: VELCADE® Plus Rituximab in Non Hodgkin's Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLLREC3
Record Dates: First submitted 2010-12-28; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Non Hodgkin's Follicular Lymphoma
Keywords: Non Hodgkin's Follicular Lymphoma; relapsed; progressed
MeSH Terms: conditions — Recurrence | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib + Rituximab (Experimental): Single arm. Patients will be treated with Bortezomib, 1,3 mg/m2 intravenous bolus (over 3-5 seconds) on days 1, 4, 8, 11 of 21 day cycle for 6 cycles and Rituximab 375 mg/m2 intravenous infusion on day 1 of cycle III, IV, V, VI. Two additional doses will be administered at week + 3 and week + 6 after cycle VI.
  Interventions: Drug: Bortezomib (VELCADE); Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib (VELCADE) — 1,3 mg/m2, intravenous bolus (over 3-5 seconds) on days 1, 4, 8, 11 of each 21 day cycle. Number of Cycles: 6.
  Other Names: VELCADE
Drug: Rituximab — 375 mg/m2 as intravenous infusion on day 1 of cycle III, IV, V, VI. Two additional doses will be administered at week + 3 and week + 6 after cycle VI.
  Other Names: Mabthera

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of the combination of Velcade and Rituximab in patients with relapsed Non Hodgkin's Follicular Lymphoma.

DETAILED DESCRIPTION:
Eligible patients will receive the combination Velcade-rituximab for up to a total of 6 cycles of Velcade and 6 infusion of rituximab.

Patients will be evaluated for clinical, laboratory, imaging parameters at baseline, during study treatment, at the end of the treatment and during follow up (every 6 months for 3 years). In the first stage, 17 patients will be treated. An interim analysis will be performed after recruitment of the first 17 evaluable patients. Aim of this analysis is to determine preliminary the activity of the treatment.If > 7 responses are observed, the accrual is continued and 24 additional patients are treated up to a total of 41. If ≤ 21 respond, the treatment is rejected as ineffective. If 22 or more respond, the treatment is judged promising for further development.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* diagnosis of relapsed or progressed disease pretreated with no more than three prior chemotherapy regimen and/or immunochemotherapy;
* age > 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* no evidence of transformation to a high grade lymphoma;
* active disease requiring treatment;
* two-dimensionally measurable disease in at least one site or evaluable disease;
* Velcade® naïve;
* life expectancy >6 months;
* no prior chemotherapy, immunotherapy or radiotherapy in the last 8 weeks;
* adequate renal function (calculated or measured creatinine clearance > 30 mL/minute), liver function aspartate aminotransferase (ASAT)/alanine aminotransferase (ALAT) < 3.0 x upper normal, total bilirubin < 2,5 x upper normal), unless due to lymphoma involvement;
* left ventricular ejection fraction (LVEF) > 50%;
* no evidence of active opportunistic infections;
* HbsAg, and hepatitis C virus (HCV) e HIV negativity. Positive serology for hepatitis B virus (HBV) and HCV admitted only upon negativity of HBV-DNA and HCV-RNA tests;
* no serious medical illness likely to interfere with participation in this clinically study;
* voluntary Written Informed Consent before performance of any study-related procedures;
* patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in validated translations. Inability (illiteracy, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible; 17. female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study;

Exclusion Criteria:

* prior diagnosis of neoplasm (except than follicular lymphoma) within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non melanomatous skin cancer;
* refractory disease (non responding patient to previous treatment);
* other investigational drug within 28 days before enrollment;
* evidence of symptomatic central nervous system (CNS) disease;
* severe impairment of bone marrow function (Absolute Neutrophil Count (ANC) < 1.5 x 109/L, platelet (PLT) < 50 x109/L within 14 days before enrollment), unless due to lymphoma involvement;
* evidence of ≥ grade 2 neuropathy within 14 days before enrollment;
* known hypersensitivity to bortezomib, boron or mannitol;
* known hypersensitivity or anaphylactic reactions to murine antibodies or proteins;
* uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 7, NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis;
* pregnant or lactating status, confirmation that the subject is no pregnant must be established by a negative serum human chorionic gonadotropin (hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post menopausal or surgically sterilized women;
* any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule; those conditions should be discussed with the patient before registration in the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Antitumor activity after complete treatment | 30 days after the last infusion of rituximab
  Evaluate the antitumor activity in terms of clinical and molecular Overall Response Rate (ORR) after 6 courses of Velcade + Rituximab followed by two additional doses of Rituximab alone

SECONDARY OUTCOMES:
Number of patients with adverse events | From start of treatment until the end of follow up period (three years)
  Evaluate the safety on the basis of recorded toxicities graded on a scale of 1 to 5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Antitumor activity after 2 cycles of Velcade alone | between 1 and 2 weeks after the end of cycle II of Velcade
  Early evaluate the antitumor activity in terms of clinical and molecular ORR after the first two cycles of therapy with Velcade® alone

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Sacchi, MD, Principal Investigator — Gruppo Italiano Studio Linfomi
Locations (1):
- Gruppo Italiano Studio Linfomi, Modena, Modena, Italy